CLINICAL TRIAL: NCT06650384
Title: Evaluation of the Efficacy and Safety of N-Acetylcysteine Versus Alpha-Lipoic Acid on the Occurrence and Severity of Colistin-Induced Nephrotoxicity in Critically Ill Patients
Brief Title: Efficacy and Safety of N-Acetylcysteine Versus Alpha-Lipoic Acid in Colistin-Induced Nephrotoxicity
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina hussein ahmed eladly, Senior Clinical Pharmacist (Principal investigator), Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RHDIRB2020110301 REC#266
Record Dates: First submitted 2024-10-13; First posted 2024-10-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Nephrotoxicity
Keywords: N-Acetylcysteine; Alpha-Lipoic Acid; Colistin; Nephrotoxicity

STUDY DESIGN:
Intervention Model Description: This study will be a prospective randomized controlled clinical trial Eligible patients will be randomly assigned by a 1:1:1 ratio using a computer-generated sequence to any of the 3 groups Group1 (n=60): colistin Group2 (n=60): colistin and N-Acetylcysteine Group3 (n=60): colistin and Alpha-lipoic acid
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (1): colistin only (No Intervention): Group1 (n=60): will receive (IV) colistin 300 mg CBA loading dose, followed 12 hours later by a maintenance dose of 150-180 mg CBA twice daily based on Crcl calculated using Cockcroft -Gault equation .
- Group(2): colistin and N-Acetylcysteine (Experimental): Group2 (n=60): will receive (IV) colistin 300mg CBA loading dose followed by a maintenance dose of 150-180 mg CBA twice daily based on Crcl calculated using Cockcroft -Gault equation in addition to enteral sachets of N-acetyl cysteine 1200 mg twice/day (acetylcysteine 600mg sachets produced by South Egypt Drug Industries Company, SEDICO)
  Interventions: Drug: Addition of sachets of N-acetyl cysteine 1200 mg twice/day to the maintenance dose of colistin
- Group(3): colistin and Alpha-lipoic acid (Experimental): Group3 (n=60): will receive (IV) colistin 300mg CBA loading dose followed by a maintenance dose 150-180 mg CBA twice daily based on Crcl calculated using Cockcroft -Gault equation in addition to enteral Alpha-lipoic acid 600mg twice daily (thiotacid 600mg produced by EVA PHARM) before meals .
  Interventions: Drug: Addition of Alpha-lipoic acid 600mg twice daily to the maintenance dose of colistin

INTERVENTIONS:
Drug: Addition of sachets of N-acetyl cysteine 1200 mg twice/day to the maintenance dose of colistin — Group2 (n=60): (IV) colistin 300mg CBA loading dose then maintenance dose of 150-180 mg CBA twice daily based on Crcl calculated using Cockcroft -Gault equation in addition to enteral sachets of N-acetyl cysteine 1200 mg twice /day
  Other Names: Acetylcysteine ® ;South Egypt Drug Industries Company, SEDICO,Egypt
  Arms: Group(2): colistin and N-Acetylcysteine
Drug: Addition of Alpha-lipoic acid 600mg twice daily to the maintenance dose of colistin — Group3 (n=60): (IV) colistin 300mg CBA loading dose then maintenance dose 150-180 mg CBA twice daily based on Crcl calculated using Cockcroft -Gault equation in addition to enteral Alpha-lipoic acid 600mg twice/day
  Other Names: Thiotacid ® ; EVA PHARM,Egypt
  Arms: Group(3): colistin and Alpha-lipoic acid

SUMMARY:
Healthcare- associated infections that caused by multi-drug-resistant Gram-negative bacteria (MDR G-ve) represent the most important problem that face the critically ill patients in the ICU. The available broad-spectrum antibiotics as penicillin, fluoroquinolones, aminoglycosides, and β-lactams fail to overcome these aggressive organisms. Accordingly, this led to the reconsideration of old drugs such as polymyxin B and polymyxin E (also known as colistin) that were previously considered to be too toxic for clinical use in the treatment of MDR G-ve bacteria. Colistin can be used as monotherapy or in combination with other antibiotics as high dose tigecycline, carbapenem or high-dose ampicillin/sulbactam.

Colistin associated acute kidney injury (CA-AKI) is the frequently observed side effect in ICU patients treated with colistin that may lead to cessation of treatment. Accordingly, it is important to monitor renal functions prior to and during colistin treatment to detect the early signs of renal injury and minimize long term renal dysfunction.

Inflammation with release of reactive oxygen species (ROS) can lead to renal tubular cells apoptosis. Several animal studies proved the beneficial effect of the concomitant use of antioxidants as N-acetylcysteine, alpha lipoic acid in preventing or attenuating colistin induced nephrotoxicity by their potent antioxidant effects Therefore, a clinical trial will be carried out to evaluate the efficacy and safety of N-acetylcysteine versus Alpha-lipoic acid in the prevention of colistin-induced nephrotoxicity in critically ill patients.

DETAILED DESCRIPTION:
Nosocomial infections caused by multi-drug-resistant Gram-negative bacteria (MDR G-ve) bacteria, particularly Acinetobacter baumannii, Pseudomonas aeruginosa and Klebsiella pneumonia represent a crucial rapidly increasing health problem worldwide nowadays.

The available effective antibiotics, including broad-spectrum penicillin, fluoroquinolones, aminoglycosides, and β-lactams (carbapenems, monobactam, and cephalosporins) often fail to combat these organisms and the pharmaceutical pipeline is still facing the problem of lack of new moieties. The new and potent β-lactam/ β-lactamase combinations antibiotics "Tigecycline and other newer highly expensive β-lactam/ β-lactamase combinations as ceftazidime/avibactam, meropenem/vaborbactam "have their concerns related to their high cost and unavailability in all countries. Moreover, they are ineffective against Metallo-β-lactamase-producing CRE. Accordingly, this led to the reconsideration of old drugs such as polymyxin B and polymyxin E (also known as colistin) that were previously considered to be too toxic for clinical use in the treatment of MDR G-ve bacteria Colistin has re-emerged for treatment of severe infections caused by multidrug-resistant Gram-negative bacteria especially Pseudomonas aeruginosa, Acinetobacter baummannii, Klebsiella pneumonia and Enterobacterales .Colistin monotherapy or colistin based synergistic combinations with a carbapenem, high-dose ampicillin/sulbactam or high dose tigecycline represent the last resort option to overcome CR-GNB in critically ill patients. Colistin (colistimethate sodium) is the inactive prodrug that is hydrolyzed to colistin that act as a cationic detergent and disrupt the bacterial cytoplasmic membrane resulting in leak of intracellular substances and cell death.

Colistin associated acute kidney injury (CA-AKI) is frequently observed in the intensive care unit (ICU) patients treated with colistin especially in patients with advanced age, other comorbidities, baseline renal dysfunction and hemodynamically unstable patients Colistin is primarily eliminated renally and may induce acute kidney injury at a rate of up to 53% Many studies have discussed the prevalence of colistin induced nephrotoxicity. One recent study in 2023 stated that the incidence of nephrotoxicity was 44.9% (95% CI; 37% to 53%) and its severity according to Kidney Disease Improving Global Outcomes (KDIGO) guidelines in 2012 was stage1 (47%), stage2 (21%) and stage3 (31%). Accordingly, it is important to monitor renal functions prior to and during colistin treatment to detect the early signs of renal injury and minimize long term renal dysfunction. A serum creatinine (SCr) is commonly used for estimation of renal function.

Cockcroft-Gault equation is the most common formula for determining creatinine clearance which estimates glomerular filtration rate (GFR). Although creatinine clearance may over-estimate GFR by (10-20%) but still remains the standard for drug dosing adjustments.

Accordingly, it is important to monitor renal functions prior to and during colistin treatment to detect the early signs of renal injury.

Inflammation with the release of many cytokines into the renal tubular cells, oxidative stress, the increased release of reactive oxygen species (ROS). Also, excessive free radical production and low antioxidant level which lead to renal tubular cells apoptosis with an effect on the mitochondria as a primary site of damage.

Mechanism of colistin induced nephrotoxicity is similar to that of contrast induced nephrotoxicity, the nephrotoxic effect of methotrexate/cisplatin (MTX/CPT) and vancomycin induced nephrotoxicity.

In several animal studies, the concomitant use of antioxidants as N-acetylcysteine, alpha lipoic acid, vitamin E, melatonin and ascorbic acid with colistin have shown promising results in preventing or attenuating colistin induced nephrotoxicity by their potent antioxidant effects that decrease ROS levels and cellular apoptosis.

NAC acts as a glutathione precursor that plays an important role in increasing the glutathione S- transferase activity that decrease the oxidative stress by neutralizing ROS Animal studies found that N-Acetylcysteine seems to have a beneficial role in the restoration of the oxidant injury caused by colistin and prevention of colistin-induced nephrotoxicity by its antioxidant effect. Nevertheless, one clinical study stated that N-Acetylcysteine 1200 mg /day did not have any effect on the prevention of colistin-induced nephrotoxicity. Double dose of N-acetylcysteine (1200 mg orally twice daily) seemed to be more effective than the standard dose (600 mg orally twice daily) in preventing contrast agent associated nephrotoxicity.

Also, the efficacy of NAC in the prevention of vancomycin induced nephrotoxicity was shown in a randomized controlled clinical trial in 2020.The mechanism of colistin induced nephrotoxicity is similar to that of contrast and vancomycin Alpha-lipoic acid (ALA) known as thioctic acid "600 mg twice daily "is an organosulfur compound found in the mitochondria. It is necessary for many enzymatic functions and can prevent nephrotoxicity through its strong antioxidant properties that act as a free radical scavenger and regenerator of endogenous antioxidants. Up till now, only one study on rats have demonstrated that ALA is an effective strategy for alleviation of colistin induced nephrotoxicity by its strong antioxidant effect.

An animal study on rats proved that the potent antioxidant, Alpha-lipoic acid (10mg/kg), attenuated nephrotoxicity induced by MTX/CPT by enhancing the activities of mitochondrial enzymes and decreasing levels of reactive oxygen species. The mechanism of colistin induced nephrotoxicity is similar to that of methotrexate/cisplatin.

Objectives: To evaluate the efficacy and safety of high dose N-acetylcysteine versus alpha-lipoic acid on the occurrence and severity of colistin-induced nephrotoxicity in critically ill patients by assessment of the following:

1. Efficacy parameters:

   * Occurrence and severity of nephrotoxicity
   * Clinical outcomes (ICU stay, mortality, dose modification and need for dialysis)
2. Safety parameters:

   * Occurrence of ARDs Methodology
   * As per our protocol, critically ill patients ≥ 18 years presenting to the critical care medicine Department-Cairo University Hospitals and initiating treatment with colistin for suspected or confirmed multi-drug-resistant Gram-negative bacterial infection (per culture) will be recruited.

     180 Eligible patients will be randomly assigned by a 1:1:1 ratio using a computer-generated sequence to any of the following 3 groups:
   * Group1 (n=60): will receive (IV) colistin 300 mg CBA loading dose, followed 12 hours later by a maintenance dose of 150-180 mg CBA twice daily based on Crcl calculated using Cockcroft -Gault equation . - Group2 (n=60): will receive (IV) colistin 300mg CBA loading dose followed by a maintenance dose of 150-180 mg CBA twice daily based on Crcl calculated using Cockcroft -Gault equation in addition to enteral sachets of N-acetyl cysteine 1200 mg twice/day (acetylcysteine 600mg sachets produced by South Egypt Drug Industries Company, SEDICO).
   * Group3 (n=60): will receive (IV) colistin 300mg CBA loading dose followed by a maintenance dose 150-180 mg CBA twice daily based on Crcl calculated using Cockcroft -Gault equation in addition to enteral Alpha-lipoic acid 600mg twice daily (thiotacid 600mg produced by EVA PHARM) before meals.

Every patient in the study will be subjected to the following:

1. Data collection

Data will be collected at baseline and at regular intervals from patient's medical files for all groups and this includes:

1. Patients demographic (gender, age, weight), Histories (social, medications) and pre-existing comorbid conditions and source of infection.

b. Severity scores for illness evaluation (baseline and at the end) "Acute Physiology and Chronic Health Evaluation II (APACHE II score), Sequential Organ Failure Assessment (SOFA score)" c- All culture results and susceptibilities. d-The use of other potentially nephrotoxic drugs will be recorded 2- Laboratory evaluation will be done initially and every other day up to the end of the duration of colistin treatment in the 3 groups for the following: Complete blood count (CBC) including total leucocytic count (TLC), hemoglobin (Hgb), platelets (PLT) count, inflammatory markers (C- reactive protein), urine output (UOP), renal functions BUN, SCr , Crcl that can be predicted from serum creatinine value using Cockcroft-Gault equation.

3- Vital signs assessments including (blood pressure, heart rate, temperature) at baseline and every other day till the end of colistin therapy 4- Clinical outcomes evaluation

-Assessment of Colistin Induced nephrotoxicity

All patients in the 3 groups will be assessed daily for the occurrence and severity of colistin induced nephrotoxicity defined by the KIDIGO, 2012 as:

Definition of Colistin induced Nephrotoxicity according to KDIGO staging (2012).

Moreover, the following will be reported for all patients:

- Average dose of colistin used daily during the duration of its use. Average duration of colistin use according to the type of infection and the clinical response.

-Other clinical outcomes: 5. Total length of ICU stays 6. Need for dose modification according to creatinine clearance 7. Need for hemodialysis 8. Mortality 4. Safety assessment: All adverse drug reactions will be monitored and reported for the 3 groups

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years
2. Critically ill patients initiating treatment with colistin for suspected or confirmed multi-drug-resistant Gram-negative bacterial infection as per culture

Exclusion Criteria:

1. Patient is in AKI according to KDIGO guidelines in 2012 KDIGO.org. Accessed at 17/2/2024)
2. Any kidney disorder including (glomerulonephritis, polycystic kidney disease, kidney stones, interstitial nephritis, renal artery stenosis and renal carcinoma).
3. Known allergy to colistin, N-acetylcysteine or alpha-lipoic acid
4. Patients with factors requiring NPO (nothing per oral)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of colistin induced nephrotoxicity | Starting from randomization date till patient ICU discharge, death from any cause or colistin discontinuation, whichever comes first, up to 14 days
  Serum creatinine of patients will be followed up daily and calculation of creatinine clearance daily during colistin/ colistin and interventional drug use in the ICU

SECONDARY OUTCOMES:
Need for dose modification or hemodialysis | Starting from randomization date till patient ICU discharge, death from any cause or colistin discontinuation, whichever comes first, up to 14 days
  All patients will be followed up daily for the need of dose adjustment or hemodialysis according to creatinine clearance calculated from the value of serum creatinine that was measured daily
Mortality | Starting from randomization date till patient ICU discharge, death from any cause, whichever comes first, up to 30 days
  Measure if patient will die or discharge from the ICU
Length of ICU stay from the start of colistin / colistin and interventional drug | Starting from randomization date till patient ICU discharge, death from any cause, whichever comes first, up to 30 days
  Measure duration of ICU stay starting from colistin/colistin and interventional drug initiation
Total duration of ICU stay | Starting from ICU admission till patient ICU discharge, death from any cause, whichever comes first, up to 90 days
  Measure of the total duration of patient stay in ICU
Incidence and frequency of occurrence of interventional drugs adverse events | Starting from addition of the interventional drugs to colistin till patient ICU discharge, death from any cause or colistin discontinuation, whichever comes first, assessed up to 14 days
  Record the incidence and number of occurrence of the adverse drug reactions of the interventional drugs ( N-acetyl cysteine or Alpha-lipoic acid)
  * Adverse events of N-acetylcysteine including nausea, vomiting, non-immune anaphylaxis that include (skin rash, flushing, bronchospasm, respiratory distress, angioedema hypotension) .
  * Adverse events of alpha lipoic acid including anorexia, arthralgia, myalgia, neuralgia, paresthesia, seizures, cough and nasopharyngitis

CONTACTS AND LOCATIONS:
Overall Officials: Dina H El Adly, MSc, Principal Investigator — Critical Care Medicine Department, Cairo University Hospitals, Cairo, Egypt; Lamia M El Wakeel, PhD, Study Director — Department of Clinical Pharmacy, Faculty of Pharmacy, Ain Shams University,Cairo, Egypt
Locations (1):
- Critical Care Medicine Department,Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aslan AT, Akova M. The Role of Colistin in the Era of New beta-Lactam/beta-Lactamase Inhibitor Combinations. Antibiotics (Basel). 2022 Feb 20;11(2):277. doi: 10.3390/antibiotics11020277. PMID 35203879
- [Background] Alshaya AI, Bin Saleh K, Aldhaeefi M, Baderldin HA, Alamody FO, Alhamdan QA, Almusallam MA, Alshaya O, Al Sulaiman K, Alshareef S, Alowais SA, Al Harbi SA, Alghamdi G. Colistin Loading Dose in Septic Patients with Gram Negative Infections. Infect Drug Resist. 2022 Apr 24;15:2159-2166. doi: 10.2147/IDR.S361244. eCollection 2022. PMID 35498632
- [Background] Assimakopoulos SF, Karamouzos V, Lefkaditi A, Sklavou C, Kolonitsiou F, Christofidou M, Fligou F, Gogos C, Marangos M. Triple combination therapy with high-dose ampicillin/sulbactam, high-dose tigecycline and colistin in the treatment of ventilator-associated pneumonia caused by pan-drug resistant Acinetobacter baumannii: a case series study. Infez Med. 2019 Mar 1;27(1):11-16. PMID 30882373
- [Background] Al-Abdulkarim DA, Alzuwayed OA, Al Ammari M, Al Halwan S, Al Maklafi N, Thomas A. Colistin-induced Nephrotoxicity in a Tertiary Teaching Hospital. Saudi J Kidney Dis Transpl. 2020 Sep-Oct;31(5):1057-1061. doi: 10.4103/1319-2442.301171. PMID 33229769
- [Background] Badri S, Soltani R, Sayadi M, Khorvash F, Meidani M, Taheri S. Effect of N-acetylcysteine against Vancomycin-Induced Nephrotoxicity: A Randomized Controlled Clinical Trial. Arch Iran Med. 2020 Jun 1;23(6):397-402. doi: 10.34172/aim.2020.33. PMID 32536177
- [Background] Bialvaei AZ, Samadi Kafil H. Colistin, mechanisms and prevalence of resistance. Curr Med Res Opin. 2015 Apr;31(4):707-21. doi: 10.1185/03007995.2015.1018989. Epub 2015 Mar 19. PMID 25697677
- [Background] Briguori C, Colombo A, Violante A, Balestrieri P, Manganelli F, Paolo Elia P, Golia B, Lepore S, Riviezzo G, Scarpato P, Focaccio A, Librera M, Bonizzoni E, Ricciardelli B. Standard vs double dose of N-acetylcysteine to prevent contrast agent associated nephrotoxicity. Eur Heart J. 2004 Feb;25(3):206-11. doi: 10.1016/j.ehj.2003.11.016. PMID 14972420
- [Background] Brown DL, Masselink AJ, Lalla CD. Functional range of creatinine clearance for renal drug dosing: a practical solution to the controversy of which weight to use in the Cockcroft-Gault equation. Ann Pharmacother. 2013 Jul-Aug;47(7-8):1039-44. doi: 10.1345/aph.1S176. Epub 2013 Jun 11. PMID 23757387
- [Background] Cakir T, Polat C, Basturk A, Gul M, Aslaner A, Durgut H, Sehirli AO, Aykac A, Bahar L, Sabuncuoglu MZ. The effect of alpha lipoic acid on rat kidneys in methotrexate induced oxidative injury. Eur Rev Med Pharmacol Sci. 2015;19(11):2132-9. PMID 26125279
- [Background] Cakirlar FK, Ciftci IH, Gonullu N. OXA-type Carbapenemases and Susceptibility of Colistin and Tigecycline Among Carbapenem-Resistant Acinetobacter Baumannii Isolates from Patients with Bacteremia in Turkey. Clin Lab. 2015;61(7):741-7. doi: 10.7754/clin.lab.2014.141116. PMID 26299073
- [Background] Ceylan B, Ozansoy M, Kilic U, Yozgat Y, Ercan C, Yildiz P, Aslan T. N-acetylcysteine suppresses colistimethate sodium-induced nephrotoxicity via activation of SOD2, eNOS, and MMP3 protein expressions. Ren Fail. 2018 Nov;40(1):423-434. doi: 10.1080/0886022X.2018.1489286. PMID 30035652
- [Background] Chien HT, Lin YC, Sheu CC, Hsieh KP, Chang JS. Is colistin-associated acute kidney injury clinically important in adults? A systematic review and meta-analysis. Int J Antimicrob Agents. 2020 Mar;55(3):105889. doi: 10.1016/j.ijantimicag.2020.105889. Epub 2020 Jan 8. PMID 31923573
- [Background] Dai C, Tang S, Velkov T, Xiao X. Colistin-Induced Apoptosis of Neuroblastoma-2a Cells Involves the Generation of Reactive Oxygen Species, Mitochondrial Dysfunction, and Autophagy. Mol Neurobiol. 2016 Sep;53(7):4685-700. doi: 10.1007/s12035-015-9396-7. Epub 2015 Aug 28. PMID 26316077
- [Background] Dalfino L, Puntillo F, Mosca A, Monno R, Spada ML, Coppolecchia S, Miragliotta G, Bruno F, Brienza N. High-dose, extended-interval colistin administration in critically ill patients: is this the right dosing strategy? A preliminary study. Clin Infect Dis. 2012 Jun;54(12):1720-6. doi: 10.1093/cid/cis286. Epub 2012 Mar 15. PMID 22423120
- [Background] Eljaaly K, Bidell MR, Gandhi RG, Alshehri S, Enani MA, Al-Jedai A, Lee TC. Colistin Nephrotoxicity: Meta-Analysis of Randomized Controlled Trials. Open Forum Infect Dis. 2021 Jan 21;8(2):ofab026. doi: 10.1093/ofid/ofab026. eCollection 2021 Feb. PMID 33623807
- [Background] El-Sayed Ahmed MAE, Zhong LL, Shen C, Yang Y, Doi Y, Tian GB. Colistin and its role in the Era of antibiotic resistance: an extended review (2000-2019). Emerg Microbes Infect. 2020 Dec;9(1):868-885. doi: 10.1080/22221751.2020.1754133. PMID 32284036
- [Background] Epperson LC, Weiss ST, Cao DJ. A Case Report of a Severe, Unusually Delayed Anaphylactoid Reaction to Intravenous N-Acetylcysteine During Treatment of Acute Acetaminophen Toxicity in an Adolescent. J Med Toxicol. 2021 Jan;17(1):75-79. doi: 10.1007/s13181-020-00804-5. Epub 2020 Aug 21. PMID 32821982
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Gai Z, Samodelov SL, Kullak-Ublick GA, Visentin M. Molecular Mechanisms of Colistin-Induced Nephrotoxicity. Molecules. 2019 Feb 12;24(3):653. doi: 10.3390/molecules24030653. PMID 30759858
- [Background] Garnacho-Montero J, Amaya-Villar R, Ferrandiz-Millon C, Diaz-Martin A, Lopez-Sanchez JM, Gutierrez-Pizarraya A. Optimum treatment strategies for carbapenem-resistant Acinetobacter baumannii bacteremia. Expert Rev Anti Infect Ther. 2015 Jun;13(6):769-77. doi: 10.1586/14787210.2015.1032254. Epub 2015 Apr 12. PMID 25865094
- [Background] Giamarellou H, Poulakou G. Multidrug-resistant Gram-negative infections: what are the treatment options? Drugs. 2009 Oct 1;69(14):1879-901. doi: 10.2165/11315690-000000000-00000. PMID 19747006
- [Background] Gunay E, Kaya S, Baysal B, Yuksel E, Arac E. Evaluation of prognosis and nephrotoxicity in patients treated with colistin in intensive care unit. Ren Fail. 2020 Nov;42(1):704-709. doi: 10.1080/0886022X.2020.1795878. PMID 32703065
- [Background] Gupta S, Portales-Castillo I, Daher A, Kitchlu A. Conventional Chemotherapy Nephrotoxicity. Adv Chronic Kidney Dis. 2021 Sep;28(5):402-414.e1. doi: 10.1053/j.ackd.2021.08.001. PMID 35190107
- [Background] Gyuraszova M, Gurecka R, Babickova J, Tothova L. Oxidative Stress in the Pathophysiology of Kidney Disease: Implications for Noninvasive Monitoring and Identification of Biomarkers. Oxid Med Cell Longev. 2020 Jan 23;2020:5478708. doi: 10.1155/2020/5478708. eCollection 2020. PMID 32082479
- [Background] Heil EL, Bork JT, Abbo LM, Barlam TF, Cosgrove SE, Davis A, Ha DR, Jenkins TC, Kaye KS, Lewis JS 2nd, Ortwine JK, Pogue JM, Spivak ES, Stevens MP, Vaezi L, Tamma PD. Optimizing the Management of Uncomplicated Gram-Negative Bloodstream Infections: Consensus Guidance Using a Modified Delphi Process. Open Forum Infect Dis. 2021 Oct 11;8(10):ofab434. doi: 10.1093/ofid/ofab434. eCollection 2021 Oct. PMID 34738022
- [Background] Hu Q, Chen J, Sun S, Deng S. Mortality-Related Risk Factors and Novel Antimicrobial Regimens for Carbapenem-Resistant Enterobacteriaceae Infections: A Systematic Review. Infect Drug Resist. 2022 Nov 28;15:6907-6926. doi: 10.2147/IDR.S390635. eCollection 2022. PMID 36465807
- [Background] Ibrahim ME. Prevalence of Acinetobacter baumannii in Saudi Arabia: risk factors, antimicrobial resistance patterns and mechanisms of carbapenem resistance. Ann Clin Microbiol Antimicrob. 2019 Jan 3;18(1):1. doi: 10.1186/s12941-018-0301-x. PMID 30606201
- [Background] Inchai J, Liwsrisakun C, Theerakittikul T, Chaiwarith R, Khositsakulchai W, Pothirat C. Risk factors of multidrug-resistant, extensively drug-resistant and pandrug-resistant Acinetobacter baumannii ventilator-associated pneumonia in a Medical Intensive Care Unit of University Hospital in Thailand. J Infect Chemother. 2015 Aug;21(8):570-4. doi: 10.1016/j.jiac.2015.04.010. Epub 2015 May 7. PMID 26026660
- [Background] Jafari F, Elyasi S. Prevention of colistin induced nephrotoxicity: a review of preclinical and clinical data. Expert Rev Clin Pharmacol. 2021 Sep;14(9):1113-1131. doi: 10.1080/17512433.2021.1933436. Epub 2021 Jun 9. PMID 34015235
- [Background] Jin J, Zhu J, Zhu Z, Kim WY, O'Rourke J, Lin Z, Chen M. Clinical efficacy and nephrotoxicity of intravenous colistin sulfate in the treatment of carbapenem-resistant gram-negative bacterial infections: a retrospective cohort study. Ann Transl Med. 2022 Oct;10(20):1137. doi: 10.21037/atm-22-4959. PMID 36388829
- [Background] Kalil AC, Metersky ML, Klompas M, Muscedere J, Sweeney DA, Palmer LB, Napolitano LM, O'Grady NP, Bartlett JG, Carratala J, El Solh AA, Ewig S, Fey PD, File TM Jr, Restrepo MI, Roberts JA, Waterer GW, Cruse P, Knight SL, Brozek JL. Management of Adults With Hospital-acquired and Ventilator-associated Pneumonia: 2016 Clinical Practice Guidelines by the Infectious Diseases Society of America and the American Thoracic Society. Clin Infect Dis. 2016 Sep 1;63(5):e61-e111. doi: 10.1093/cid/ciw353. Epub 2016 Jul 14. PMID 27418577
- [Background] Kengkla K, Kongpakwattana K, Saokaew S, Apisarnthanarak A, Chaiyakunapruk N. Comparative efficacy and safety of treatment options for MDR and XDR Acinetobacter baumannii infections: a systematic review and network meta-analysis. J Antimicrob Chemother. 2018 Jan 1;73(1):22-32. doi: 10.1093/jac/dkx368. PMID 29069421
- [Background] Kilic I, Ayar Y, Ceylan I, Kaya PK, Caliskan G. Nephrotoxicity caused by colistin use in ICU: a single centre experience. BMC Nephrol. 2023 Oct 13;24(1):302. doi: 10.1186/s12882-023-03334-8. PMID 37833622
- [Background] Larki RA, Jamali B, Meidani M, Mousavi S. Serum Cystatin C for Evaluation of Acute Kidney Injury in Adults Treated with Colistin. J Res Pharm Pract. 2018 Oct-Dec;7(4):178-181. doi: 10.4103/jrpp.JRPP_18_53. PMID 30622984
- [Background] Lee YM, Bae SY, Won NH, Pyo HJ, Kwon YJ. Alpha-lipoic acid attenuates cisplatin-induced tubulointerstitial injuries through inhibition of mitochondrial bax translocation in rats. Nephron Exp Nephrol. 2009;113(4):e104-12. doi: 10.1159/000235754. Epub 2009 Aug 27. PMID 19713707
- [Background] Levey AS, Perrone RD, Madias NE. Serum creatinine and renal function. Annu Rev Med. 1988;39:465-90. doi: 10.1146/annurev.me.39.020188.002341. PMID 3285786
- [Background] Liang CA, Lin YC, Lu PL, Chen HC, Chang HL, Sheu CC. Antibiotic strategies and clinical outcomes in critically ill patients with pneumonia caused by carbapenem-resistant Acinetobacter baumannii. Clin Microbiol Infect. 2018 Aug;24(8):908.e1-908.e7. doi: 10.1016/j.cmi.2017.10.033. Epub 2017 Nov 3. PMID 29108947
- [Background] Liu J, Shu Y, Zhu F, Feng B, Zhang Z, Liu L, Wang G. Comparative efficacy and safety of combination therapy with high-dose sulbactam or colistin with additional antibacterial agents for multiple drug-resistant and extensively drug-resistant Acinetobacter baumannii infections: A systematic review and network meta-analysis. J Glob Antimicrob Resist. 2021 Mar;24:136-147. doi: 10.1016/j.jgar.2020.08.021. Epub 2020 Sep 2. PMID 32889142
- [Background] Mazuski JE, Tessier JM, May AK, Sawyer RG, Nadler EP, Rosengart MR, Chang PK, O'Neill PJ, Mollen KP, Huston JM, Diaz JJ Jr, Prince JM. The Surgical Infection Society Revised Guidelines on the Management of Intra-Abdominal Infection. Surg Infect (Larchmt). 2017 Jan;18(1):1-76. doi: 10.1089/sur.2016.261. PMID 28085573
- [Background] Mirjalili M, Mirzaei E, Vazin A. Pharmacological agents for the prevention of colistin-induced nephrotoxicity. Eur J Med Res. 2022 May 7;27(1):64. doi: 10.1186/s40001-022-00689-w. PMID 35525994
- [Background] Modi K, Padala SA, Gupta M. Contrast-Induced Nephropathy. 2025 Jan 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK448066/ PMID 28846220
- [Background] Morgan A, Galal MK, Ogaly HA, Ibrahim MA, Abd-Elsalam RM, Noshy P. Tiron ameliorates oxidative stress and inflammation in titanium dioxide nanoparticles induced nephrotoxicity of male rats. Biomed Pharmacother. 2017 Sep;93:779-787. doi: 10.1016/j.biopha.2017.07.006. Epub 2017 Jul 12. PMID 28709131
- [Background] Mosayebi S, Soltani R, Shafiee F, Assarzadeh S, Hakamifard A. Evaluation of the Effectiveness of N-Acetylcysteine in the Prevention of Colistin-Induced Nephrotoxicity: A Randomized Controlled Clinical Trial. J Res Pharm Pract. 2022 May 25;10(4):159-165. doi: 10.4103/jrpp.jrpp_90_21. eCollection 2021 Oct-Dec. PMID 35769842
- [Background] Nang SC, Azad MAK, Velkov T, Zhou QT, Li J. Rescuing the Last-Line Polymyxins: Achievements and Challenges. Pharmacol Rev. 2021 Apr;73(2):679-728. doi: 10.1124/pharmrev.120.000020. PMID 33627412
- [Background] Nation RL, Garonzik SM, Li J, Thamlikitkul V, Giamarellos-Bourboulis EJ, Paterson DL, Turnidge JD, Forrest A, Silveira FP. Updated US and European Dose Recommendations for Intravenous Colistin: How Do They Perform? Clin Infect Dis. 2016 Mar 1;62(5):552-558. doi: 10.1093/cid/civ964. Epub 2015 Nov 25. PMID 26607424
- [Background] Nation RL, Garonzik SM, Thamlikitkul V, Giamarellos-Bourboulis EJ, Forrest A, Paterson DL, Li J, Silveira FP. Dosing guidance for intravenous colistin in critically-ill patients. Clin Infect Dis. 2017 Mar 1;64(5):565-571. doi: 10.1093/cid/ciw839. Epub 2016 Dec 23. PMID 28011614
- [Background] Nguyen H, Pellegrini MV, Gupta V. Alpha-Lipoic Acid. 2024 Jan 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK564301/ PMID 33231971
- [Background] Oktan MA, Heybeli C, Ural C, Kocak A, Bilici G, Cavdar Z, Ozbal S, Arslan S, Yilmaz O, Cavdar C. Alpha-lipoic acid alleviates colistin nephrotoxicity in rats. Hum Exp Toxicol. 2021 May;40(5):761-771. doi: 10.1177/0960327120966043. Epub 2020 Oct 28. PMID 33111558
- [Background] Ordooei Javan A, Shokouhi S, Sahraei Z. A review on colistin nephrotoxicity. Eur J Clin Pharmacol. 2015 Jul;71(7):801-10. doi: 10.1007/s00228-015-1865-4. Epub 2015 May 27. PMID 26008213
- [Background] Ozkan G, Ulusoy S, Orem A, Alkanat M, Mungan S, Yulug E, Yucesan FB. How does colistin-induced nephropathy develop and can it be treated? Antimicrob Agents Chemother. 2013 Aug;57(8):3463-9. doi: 10.1128/AAC.00343-13. Epub 2013 Apr 29. PMID 23629704
- [Background] Ozyilmaz E, Ebinc FA, Derici U, Gulbahar O, Goktas G, Elmas C, Oguzulgen IK, Sindel S. Could nephrotoxicity due to colistin be ameliorated with the use of N-acetylcysteine? Intensive Care Med. 2011 Jan;37(1):141-6. doi: 10.1007/s00134-010-2038-7. Epub 2010 Sep 16. PMID 20845026
- [Background] Plachouras D, Karvanen M, Friberg LE, Papadomichelakis E, Antoniadou A, Tsangaris I, Karaiskos I, Poulakou G, Kontopidou F, Armaganidis A, Cars O, Giamarellou H. Population pharmacokinetic analysis of colistin methanesulfonate and colistin after intravenous administration in critically ill patients with infections caused by gram-negative bacteria. Antimicrob Agents Chemother. 2009 Aug;53(8):3430-6. doi: 10.1128/AAC.01361-08. Epub 2009 May 11. PMID 19433570
- [Background] Prasannan BK, Mukthar FC, Unni VN, Mohan S, Vinodkumar K. Colistin Nephrotoxicity-Age and Baseline kidney Functions Hold the Key. Indian J Nephrol. 2021 Sep-Oct;31(5):449-453. doi: 10.4103/ijn.IJN_130_20. Epub 2021 Sep 21. PMID 34880554
- [Background] Rabi R, Enaya A, Sweileh MW, Aiesh BM, Namrouti A, Hamdan ZI, Abugaber D, Nazzal Z. Comprehensive Assessment of Colistin Induced Nephrotoxicity: Incidence, Risk Factors and Time Course. Infect Drug Resist. 2023 May 15;16:3007-3017. doi: 10.2147/IDR.S409964. eCollection 2023. PMID 37215302
- [Background] Rigatto MH, Falci DR, Zavascki AP. Clinical Use of Polymyxin B. Adv Exp Med Biol. 2019;1145:197-218. doi: 10.1007/978-3-030-16373-0_14. PMID 31364080
- [Background] Sant B, Rao PV, Nagar DP, Pant SC, Bhasker AS. Evaluation of abrin induced nephrotoxicity by using novel renal injury markers. Toxicon. 2017 Jun 1;131:20-28. doi: 10.1016/j.toxicon.2017.03.007. Epub 2017 Mar 10. PMID 28288935
- [Background] Somani SM, Husain K, Whitworth C, Trammell GL, Malafa M, Rybak LP. Dose-dependent protection by lipoic acid against cisplatin-induced nephrotoxicity in rats: antioxidant defense system. Pharmacol Toxicol. 2000 May;86(5):234-41. doi: 10.1034/j.1600-0773.2000.d01-41.x. PMID 10862506
- [Background] Tsuji BT, Pogue JM, Zavascki AP, Paul M, Daikos GL, Forrest A, Giacobbe DR, Viscoli C, Giamarellou H, Karaiskos I, Kaye D, Mouton JW, Tam VH, Thamlikitkul V, Wunderink RG, Li J, Nation RL, Kaye KS. International Consensus Guidelines for the Optimal Use of the Polymyxins: Endorsed by the American College of Clinical Pharmacy (ACCP), European Society of Clinical Microbiology and Infectious Diseases (ESCMID), Infectious Diseases Society of America (IDSA), International Society for Anti-infective Pharmacology (ISAP), Society of Critical Care Medicine (SCCM), and Society of Infectious Diseases Pharmacists (SIDP). Pharmacotherapy. 2019 Jan;39(1):10-39. doi: 10.1002/phar.2209. PMID 30710469
- [Background] Tumbarello M, Losito AR, Giamarellou H. Optimizing therapy in carbapenem-resistant Enterobacteriaceae infections. Curr Opin Infect Dis. 2018 Dec;31(6):566-577. doi: 10.1097/QCO.0000000000000493. PMID 30379732
- [Background] Tunkel AR, Hartman BJ, Kaplan SL, Kaufman BA, Roos KL, Scheld WM, Whitley RJ. Practice guidelines for the management of bacterial meningitis. Clin Infect Dis. 2004 Nov 1;39(9):1267-84. doi: 10.1086/425368. Epub 2004 Oct 6. No abstract available. PMID 15494903
- [Background] Tunkel AR, Hasbun R, Bhimraj A, Byers K, Kaplan SL, Scheld WM, van de Beek D, Bleck TP, Garton HJL, Zunt JR. 2017 Infectious Diseases Society of America's Clinical Practice Guidelines for Healthcare-Associated Ventriculitis and Meningitis. Clin Infect Dis. 2017 Mar 15;64(6):e34-e65. doi: 10.1093/cid/ciw861. PMID 28203777
- [Background] Tylicki L, Rutkowski B, Horl WH. Antioxidants: a possible role in kidney protection. Kidney Blood Press Res. 2003;26(5-6):303-14. doi: 10.1159/000073936. PMID 14610334
- [Background] Wang SH, Yang KY, Sheu CC, Chen WC, Chan MC, Feng JY, Chen CM, Wu BR, Zheng ZR, Chou YC, Peng CK; T.-CARE (Taiwan Critical Care, Infection) Group. The necessity of a loading dose when prescribing intravenous colistin in critically ill patients with CRGNB-associated pneumonia: a multi-center observational study. Crit Care. 2022 Apr 4;26(1):91. doi: 10.1186/s13054-022-03947-9. PMID 35379303
- [Background] Winter MA, Guhr KN, Berg GM. Impact of various body weights and serum creatinine concentrations on the bias and accuracy of the Cockcroft-Gault equation. Pharmacotherapy. 2012 Jul;32(7):604-12. doi: 10.1002/j.1875-9114.2012.01098.x. Epub 2012 May 10. PMID 22576791
- [Background] Yahav D, Franceschini E, Koppel F, Turjeman A, Babich T, Bitterman R, Neuberger A, Ghanem-Zoubi N, Santoro A, Eliakim-Raz N, Pertzov B, Steinmetz T, Stern A, Dickstein Y, Maroun E, Zayyad H, Bishara J, Alon D, Edel Y, Goldberg E, Venturelli C, Mussini C, Leibovici L, Paul M; Bacteremia Duration Study Group. Seven Versus 14 Days of Antibiotic Therapy for Uncomplicated Gram-negative Bacteremia: A Noninferiority Randomized Controlled Trial. Clin Infect Dis. 2019 Sep 13;69(7):1091-1098. doi: 10.1093/cid/ciy1054. PMID 30535100
- [Background] Yahav D, Giske CG, Gramatniece A, Abodakpi H, Tam VH, Leibovici L. New beta-Lactam-beta-Lactamase Inhibitor Combinations. Clin Microbiol Rev. 2020 Nov 11;34(1):e00115-20. doi: 10.1128/CMR.00115-20. Print 2020 Dec 16. PMID 33177185
- [Background] Yousef JM, Chen G, Hill PA, Nation RL, Li J. Ascorbic acid protects against the nephrotoxicity and apoptosis caused by colistin and affects its pharmacokinetics. J Antimicrob Chemother. 2012 Feb;67(2):452-9. doi: 10.1093/jac/dkr483. Epub 2011 Nov 28. PMID 22127588
- [Background] Yu SN, Kim T, Park SY, Lee YM, Park KH, Lee EJ, Jeon MH, Choo EJ, Kim TH, Lee MS, Park SY. Predictors of Acute Kidney Injury and 28-Day Mortality in Carbapenem-Resistant Acinetobacter baumannii Complex Bacteremia. Microb Drug Resist. 2021 Aug;27(8):1029-1036. doi: 10.1089/mdr.2020.0312. Epub 2021 Mar 3. PMID 33656377
- [Background] Zhang J, McCullough PA. Lipoic Acid in the Prevention of Acute Kidney Injury. Nephron. 2016;134(3):133-140. doi: 10.1159/000448666. Epub 2016 Sep 8. PMID 27603173
- See also: Hintze J. (2011).PASS11 — http://www.ncss.com/
- See also: Kidney Disease Improving Global outcome (KDIGO — http://kdigo.org/guidelines/acute-kidney-injury/